CLINICAL TRIAL: NCT06743594
Title: Effects of Laser Species and Ocular Antioxidant Activity on Postoperative Inflammation, Oxidative Stress and Visual Prognosis in Patients Undergoing Ophthalmic Surgery - a Comparative Study.
Brief Title: Measurement of Antioxidant Activity and Oxidative Stress in Patients Undergoing Ophthalmic Surgery.
Status: Recruiting | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Taipei Nobel Eye Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 202401405A3
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2024-12

CONDITIONS: Cataract; Myopia
Keywords: antioxidants
MeSH Terms: conditions — Cataract; Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — tear, aqueous humor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- LASIK: Femtosecond-LASIK in myopia
- KLEx: Kerato-lenticule Extraction in myopia
- Traditional Cataract Surgery: Cataract Surgery with Phacoemulsification
- Laser-Assisted Cataract Surgery: Cataract Surgery with LenSx Femtosecond Laser

SUMMARY:
This trial hypothesized that novel laser refractive surgery techniques (LASIK, KLEx) or laser-assisted cataract surgery (FLACAS) could suppress postoperative inflammation and improve recovery in patients by reducing oxidative stress generated by the surgical procedure. It is also intended to verify whether the new laser technology is necessary for clinical use in groups with low antioxidant activity through the detection of antioxidant activity in the eyes of patients.

DETAILED DESCRIPTION:
Simultaneously measure total reactive oxygen species (ROS), antioxidant capacity (TAC) and ascorbic acid (AA) in aqueous humor (cataract surgery only) or tears. All patients underwent the same examination at our institution, including uncorrected visual acuity (UCVA), intraocular pressure (IOP), as well as central corneal thickness (CCT) with pneumatic tonometer, apparent refraction with autorefractor, and corneal curvature with keratometer. The axial length (AXL), anterior chamber depth (ACD) and lens thickness (LT) were measured by optical biometer.

ELIGIBILITY:
Inclusion Criteria:

* at least 20 years old
* corneal refractive surgery or cataract surgery patients

Exclusion Criteria:

* patients with eye infections
* presence of severe retinal disease
* presence of severe eye injury or severe ptosis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study included patients with the following conditions: (1) at least 20 years old, (2) expected to undergo corneal refractive surgery or cataract surgery.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-03-14 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
TAC in tears at 1 week | Before the operation and 1 week after surgery.
  Change of Total Antioxidant Capacity (TAC) from Baseline to 1 week after surgery.
TAC in tears at 1 month | Before the operation and 1 month after surgery.
  Change of Total Antioxidant Capacity (TAC) from Baseline to 1 month after surgery.
TAC in tears at 2 months | Before the operation and 2 months after surgery.
  Change of Total Antioxidant Capacity (TAC) from Baseline to 2 months after surgery.
TAC in tears at 3 months | Before the operation and 3 months after surgery.
  Change of Total Antioxidant Capacity (TAC) from Baseline to 3 months after surgery.
AA in tears at 1 week | Before the operation and 1 week after surgery.
  Change of Ascorbic Acid (AA) from Baseline to 1 week after surgery.
AA in tears at 1 month | Before the operation and 1 month after surgery.
  Change of Ascorbic Acid (AA) from Baseline to 1 month after surgery.
AA in tears at 2 months | Before the operation and 2 months after surgery.
  Change of Ascorbic Acid (AA) from Baseline to 2 months after surgery.
AA in tears at 3 months | Before the operation and 3 months after surgery.
  Change of Ascorbic Acid (AA) from Baseline to 3 months after surgery.
ROS in tears at 1 week | Before the operation and 1 week after surgery.
  Change of Reactive Oxygen Species (ROS) from Baseline to 1 week after surgery.
ROS in tears at 1 month | Before the operation and 1 month after surgery.
  Change of Reactive Oxygen Species (ROS) from Baseline to 1 month after surgery.
ROS in tears at 2 months | Before the operation and 2 months after surgery.
  Change of Reactive Oxygen Species (ROS) from Baseline to 2 moths after surgery.
ROS in tears at 3 months | Before the operation and 3 months after surgery.
  Change of Reactive Oxygen Species (ROS) from Baseline to 3 months after surgery.
TAC in aqueous humor at the next day | Before the operation and one day after surgery.
  Change of Total Antioxidant Capacity (TAC) in aqueous humor from Baseline to one day after surgery
AA in aqueous humor at the next day | Before the operation and one day after surgery.
  Change of Ascorbic Acid (AA) in aqueous humor from Baseline to one day after surgery
ROS in aqueous humor at the next day | Before the operation and one day after surgery.
  Change of Reactive Oxygen Species (ROS) in aqueous humor from Baseline to one day after surgery

SECONDARY OUTCOMES:
BCVA | Before surgery
  Examination of best corrected visual acuity (BCVA)
UCVA at 1 week | 1 week after surgery
  Examination of uncorrected visual acuity (UCVA)
UCVA at 1 month | 1 month after surgery
  Examination of uncorrected visual acuity (UCVA)
UCVA at 2 months | 2 months after surgery
  Examination of uncorrected visual acuity (UCVA)
UCVA at 3 months | 3 months after surgery
  Examination of uncorrected visual acuity (UCVA)

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Taipei Nobel Eye Clinic, Taipei
  - Chang Gung Memorial Hospital, Taoyuan District

REFERENCES:
- [Background] Umapathy A, Donaldson P, Lim J. Antioxidant delivery pathways in the anterior eye. Biomed Res Int. 2013;2013:207250. doi: 10.1155/2013/207250. Epub 2013 Sep 26. PMID 24187660
- [Background] Merida S, Villar VM, Navea A, Desco C, Sancho-Tello M, Peris C, Bosch-Morell F. Imbalance Between Oxidative Stress and Growth Factors in Human High Myopia. Front Physiol. 2020 May 14;11:463. doi: 10.3389/fphys.2020.00463. eCollection 2020. PMID 32477165
- [Background] Tsao YT, Wu WC, Chen KJ, Liu CF, Hsueh YJ, Cheng CM, Chen HC. An Assessment of Cataract Severity Based on Antioxidant Status and Ascorbic Acid Levels in Aqueous Humor. Antioxidants (Basel). 2022 Feb 16;11(2):397. doi: 10.3390/antiox11020397. PMID 35204279
- [Background] Kato K, Miyake K, Hirano K, Kondo M. Management of Postoperative Inflammation and Dry Eye After Cataract Surgery. Cornea. 2019 Nov;38 Suppl 1:S25-S33. doi: 10.1097/ICO.0000000000002125. PMID 31498249
- [Background] Hsueh YJ, Meir YJ, Lai JY, Huang CC, Lu TT, Ma DH, Cheng CM, Wu WC, Chen HC. Ascorbic acid ameliorates corneal endothelial dysfunction and enhances cell proliferation via the noncanonical GLUT1-ERK axis. Biomed Pharmacother. 2021 Dec;144:112306. doi: 10.1016/j.biopha.2021.112306. Epub 2021 Oct 15. PMID 34656060
- [Background] Dong Z, Zhou X, Wu J, Zhang Z, Li T, Zhou Z, Zhang S, Li G. Small incision lenticule extraction (SMILE) and femtosecond laser LASIK: comparison of corneal wound healing and inflammation. Br J Ophthalmol. 2014 Feb;98(2):263-9. doi: 10.1136/bjophthalmol-2013-303415. Epub 2013 Nov 13. PMID 24227802
- [Background] Seen S, Tong L. Dry eye disease and oxidative stress. Acta Ophthalmol. 2018 Jun;96(4):e412-e420. doi: 10.1111/aos.13526. Epub 2017 Aug 21. PMID 28834388
- [Background] Vallabh NA, Romano V, Willoughby CE. Mitochondrial dysfunction and oxidative stress in corneal disease. Mitochondrion. 2017 Sep;36:103-113. doi: 10.1016/j.mito.2017.05.009. Epub 2017 May 23. PMID 28549842
- [Background] Wong AHY, Cheung RKY, Kua WN, Shih KC, Chan TCY, Wan KH. Dry Eyes After SMILE. Asia Pac J Ophthalmol (Phila). 2019 Sep-Oct;8(5):397-405. doi: 10.1097/01.APO.0000580136.80338.d0. PMID 31490199
- [Background] Nair S, Kaur M, Sharma N, Titiyal JS. Refractive surgery and dry eye - An update. Indian J Ophthalmol. 2023 Apr;71(4):1105-1114. doi: 10.4103/IJO.IJO_3406_22. PMID 37026241